CLINICAL TRIAL: NCT00483392
Title: Treatment of Hyperglycaemia and Insulin Resistance in HIV Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J3-3545; Slovenia grant J3-3545
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2007-06-07 (Estimated); Status verified 2007-06

CONDITIONS: Insulin Resistance
Keywords: insulin; rosiglitazone; metformin; hiv; protease inhibitors
MeSH Terms: conditions — Insulin Resistance; Acquired Immunodeficiency Syndrome | interventions — rosiglitazone-metformin combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: metformin, rosiglitazone

SUMMARY:
The purpose of this study is to evaluate and compare the effects of treatment with rosiglitazone and metformin on insulin resistance in patients infected with Human Immunodeficiency Virus on stable Highly Active Antiretroviral Therapy including a Protease Inhibitor after the period of 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* documented HIV infection
* stable Protease Inhibitor containing HAART regimen for at least 12 months
* impaired glucose tolerance
* elevated insulin levels (above 20 mIU/l)

Exclusion Criteria:

* patients already taking oral hypoglycaemic treatment or insulin
* heart failure NYHA I-IV
* liver disease or kidney disease
* elevated AST or ALT above 2 times upper normal range
* elevated creatinine (above 150 mmol/l)

Ages: 18 Years to 60 Years | Sex: Male
Age Groups: Adult

PRIMARY OUTCOMES:
fasting plasma glucose, basal insulin levels | 48 weeks

SECONDARY OUTCOMES:
insulin resistance, beta cell function | 48 week

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Janez, MD, PhD, Study Chair — Department of Endocrinology, Diabetes and Metabolic Diseases, Medical Center Ljubljana, Zaloska 7, 1525 Ljubljana, Slovenia
Locations (1):
- Department of Endocrinology, Diabetes and Metabolic diseases, Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Silic A, Janez A, Tomazic J, Karner P, Vidmar L, Sharma P, Maticic M. Effect of rosiglitazone and metformin on insulin resistance in patients infected with human immunodeficiency virus receiving highly active antiretroviral therapy containing protease inhibitor: randomized prospective controlled clinical trial. Croat Med J. 2007 Dec;48(6):791-9. doi: 10.3325/cmj.2007.6.791. PMID 18074413